CLINICAL TRIAL: NCT02719418
Title: Study of the Bioaccumulation of Tinzaparin in Renally Impaired Patients When Given at Prophylactic Doses
Acronym: STRIP
Status: Completed | Type: Observational
Sponsor: Maisonneuve-Rosemont Hospital (Other)
Responsible Party: Principal Investigator, Jean-Philippe Lafrance, MD., M.Sc., FRCPC, Maisonneuve-Rosemont Hospital
Other Study IDs: STRIP-001
Record Dates: First submitted 2016-03-14; First posted 2016-03-25 (Estimated); Last update posted 2018-12-13 (Actual); Status verified 2018-12

CONDITIONS: Renal Insufficiency, Chronic; Deep Venous Thrombosis, Protection Against
Keywords: Thromboembolism; Venous Thrombosis; Embolism and Thrombosis; Chronic Renal Diseases; Kidney Failure, Chronic; Renal Failure, Chronic; Venous Thromboembolism; Tinzaparin; Innohep; Heparin, Low-Molecular-Weight
MeSH Terms: conditions — Renal Insufficiency, Chronic; Venous Thrombosis; Thromboembolism; Embolism and Thrombosis; Kidney Failure, Chronic; Venous Thromboembolism | interventions — Tinzaparin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Tinzaparin: Hospitalized patients with chronic renal insufficiency (eGFR ≤ 30 mL/min/1.73 m2) at risk of VTE secondary to non-surgical reasons and receiving thromboprophylactic doses of tinzaparin 3500 or 4500 unit sub-cutaneous once daily.
  Interventions: Drug: Tinzaparin

INTERVENTIONS:
Drug: Tinzaparin — 3500 Unit or 4500 Unit subcutaneous once daily
  Other Names: Innohep

SUMMARY:
The purpose of this study is to assess if accumulation of anti-Xa activity occurs after repeated daily administration of prophylactic doses of tinzaparin in patients with severe chronic kidney disease (CKD) requiring thromboprophylaxis for non-surgical conditions.

It is anticipated that tinzaparin used at a fixed dose for thromboprophylaxis in severe CKD patients (eGFR ≤ 30 ml/min /1.73 m2) at risk for venous thromboembolism (VTE) will not bioaccumulate at a significant level, meaning an increase of ≥ 20% of the anti-Xa mean level between day 2 or 3 and day 5.

DETAILED DESCRIPTION:
STUDY DESIGN :

Prospective, monocentric, open-label, single-arm, observational cohort study

Subjects hospitalized for non-surgical reasons by medical departments (ie Nephrology, Pneumology, Cardiology and Internal medicine) with chronic kidney disease (baseline eGFR ≤30 ml/min/1.73 m2) receiving tinzaparin prophylaxis at a dose of 3500 IU (or 4500 IU if BMI > 30kg/m2) once-daily.

Pharmacokinetic parameters: Peak anti-Xa analyses done after 2 (or 3), 5, and 8 days of treatment, and one trough anti-Xa analysis on day 5. The bioaccumulation of tinzaparin will be assessed by determining whether this dosing regimen is associated with an excessive increase in anti-Xa levels over the course of the treatment (see below for statistical analysis).

RECRUITMENT PROCESS:

A systematic screening for potential study subjects will be made by the research coordinators based on key computer searches fields throughout four different softwares. Through these databases, researchers will be able to perform a preliminary selection of any of the eligible subjects by identifying hospitalized patients that will ultimately be treated. The pharmacists responsible for validation of tinzaparin prescriptions at the pharmacy department will work with the research team at the initial screening by identifying eligible candidates. Since the choice of prescribed agents is to the prescriber's discretion, the recruitment procedures will be triggered mainly as soon as a prescription of tinzaparin at thromboprophylaxic dose is written.Subjects who meet the inclusion criteria and do not meet any exclusion criteria will be considered eligible candidates and additional baseline information will be collected at that point, such as ethnicity and sex. The eligible participant will be addressed directly by a member of the research team. Informed consent will be sought and documented through the Information Form and Informed Consent (FIC) already approved by the ethics committee the hospital.

DATA COLLECTION:

Four blood samples, three of which will be collected 4±1 hours after the injection of tinzaparin at days 2 (or 3), at day 5 and at day 8, and one trough that will be collected at day 5.

Pre-identified tubes (encoded) will be provided to the nursing and the sample shipping staff with specific instructions for manipulation of the blood sample and shipping to the laboratory.

STUDY SAMPLE:

In this study, it is considered that bioaccumulation should be statistically significant if Cmax of anti-Xa are increased by at least 20%. Estimation of the population size was performed using information obtained from Mahé et al. due to the similar nature of the population studied. As for mean plasma anti-Xa peak levels, a study done by Bara L et al. showed that 431 patients receiving 3 500 IU of tinzaparin for thromboprophylaxis had a mean of 0.15 IU/ml, which is the dose that will be given to most of the subjects in the present study. Based on the coefficient variation of Mahé et al. of 0.36 and the mean plasma anti-Xa level found by Bara L. et al, a standard deviation of 0.05 IU/ml was established, considering that the same coefficient of variation should be maintained across the dose administered. For the purpose of this study, researchers presumed an identical variance between all anti-Xa levels regardless of the day of blood sample collection. According to the null hypothesis, the mean of the distribution is 0.15 IU/ml while for the alternative hypothesis; the average would be 0.18 IU/ml (since established cut-off is a 20% increase). With a paired one-tailed t test, an alpha error of 0.05, a power of 0.90, and a strong correlation between measurements (r=0.7) , 25 participants are required to detect an increase ≥ 20% in anti-Xa activity between sampling on day 2 or 3 and at maximum of 8 days.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old
* A prescription of prophylactic tinzaparin (3500 IU or 4500 IU) has been initiated by order of the treating physician
* Patient admitted for medical reasons by one (but not limited to) of the following wards: nephrology, internal medicine, cardiology or pneumology
* Chronic severe renal impairment defined as an eGFR ≤ 30 mL/min/1.73 m2 at the moment of prescription and when available, eGFR at baseline, ie ≤ 30 ml/min/1.73 m2 for the last 3 months
* Estimated length of stay ≥ 5 days
* Written informed consent obtained within at most 3 ± 1 hours after the second or third dose of tinzaparin.

Exclusion Criteria:

* Super obese (Body-mass Index (BMI) > 50kg/m2)
* Treatment with UFH, LMWH or oral factor Xa inhibitors <48h prior starting the first dose of tinzaparin
* Prophylaxis with LMWH other than tinzaparin < 48h prior starting the first dose of tinzaparin
* Prophylaxis with heparin < 12h prior starting the first dose of tinzaparin
* Treatment with argatroban, bivalirudin < 24 hours prior starting the first dose of tinzaparin
* Treatment with oral direct thrombin inhibitors, danaparoid, fondaparinux, or anti-vitamin K agents for < 7 days prior to starting the first dose of tinzaparin
* Acute renal failure in an individual with baseline eGFR > 30 ml/min/1.73 m2
* Prophylactic tinzaparin in use for more than 72h before inclusion
* Severe liver insufficiency (Child- Pugh C)
* Anuria or chronically dialysed patients (or eGFR < 5 ml/min/1.73 m2)
* Participation in another study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects with severe renal impairment (eGFR ≤ 30 mL/min/1.73 m2) at risk of VTE secondary to non-surgical reasons and receiving thromboprophylactic doses of tinzaparin. The study sample will be selected from patients that are hospitalized by medical departments (i.e. nephrology, internal medicine, cardiology, pneumology) and on the transitional hospitalization unit.
Sampling Method: Probability Sample
Enrollment: 28 (Actual)
Dates: Start 2016-02-01 (Actual); Primary Completion 2016-09-30 (Actual); Study Completion 2018-12-12 (Actual)

PRIMARY OUTCOMES:
Peak anti-Xa levels in patients with eGFR ≤ 30 mL/min/1.73 m2 receiving repeated daily doses of tinzaparin for VTE prophylaxis | 4±1 hours after administration of tinzaparin on days 2 or 3, and 5.
  To compare the anti-Xa levels between day 2 (or 3) and day 5 in order to assess if bioaccumulation occurs at a significant level, meaning an increase of ≥ 20% of the anti-Xa mean level.The anti-Xa levels will be measured 4±1 hours after administration, which corresponds to the maximal concentration (Cmax) of tinzaparin anti-Xa activity.

SECONDARY OUTCOMES:
Peak anti-Xa levels in patients with eGFR ≤ 20 mL/min/1.73 m2 receiving repeated daily doses of tinzaparin for VTE prophylaxis | 4±1 hours after administration of tinzaparin on days 2 or 3, and 5.
  To compare the anti-Xa levels between day 2 (or 3) and day 5 in order to assess if bioaccumulation occurs at a significant level, meaning an increase of ≥ 20% of the anti-Xa mean level. The anti-Xa levels will be measured 4±1 hours after administration, which corresponds to the Cmax of tinzaparin of the anti-Xa activity.
Peak anti-Xa levels in patients with eGFR ≤ 30 mL/min/1.73 m2 receiving repeated daily doses of tinzaparin for VTE prophylaxis | 4±1 hours after administration of tinzaparin on days 2 or 3, and 8.
  To compare the anti-Xa levels between day 2 (or 3) and day 8 in order to assess if bioaccumulation occurs at a significant level, meaning an increase of ≥ 20% of the anti-Xa mean level. The anti-Xa levels will be measured 4±1 hours after administration, which corresponds to the Cmax of tinzaparin anti-Xa activity.
Anti-Xa trough level | On day 5
  To explore the safety of tinzaparin at daily prophylactic doses for VTE in renally impaired patients by measuring the trough anti-Xa level (Cmin) on day 5, and to assess the proportion of participants with a trough above 0.40 IU/mL. A level of just above 0.50 IU/ml anti-Xa activity (close to 0.4 IU/ml) is within the range of therapeutic anticoagulation for the treatment of VTE with tinzaparin and, therefore, is considered excessive anticoagulation for VTE prophylaxis.

OTHER OUTCOMES:
Bleeding events or thrombotic events | From time of entry in the study to end of study (maximum of 8 days)
  To document the incidence of the following clinical events: non major clinically relevant bleeding events, major bleeding events and VTE (symptomatic or not) in study participants during the time that they are under study.

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Philippe Lafrance, Principal Investigator — Maisonneuve-Rosemont Hospital
Locations (1):
- Maisonneuve-Rosemont Hospital, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Turpie AG, Leizorovicz A. Prevention of venous thromboembolism in medically ill patients: a clinical update. Postgrad Med J. 2006 Dec;82(974):806-9. doi: 10.1136/pgmj.2005.044107. PMID 17148703
- [Background] Goldhaber SZ, Dunn K, MacDougall RC. New onset of venous thromboembolism among hospitalized patients at Brigham and Women's Hospital is caused more often by prophylaxis failure than by withholding treatment. Chest. 2000 Dec;118(6):1680-4. doi: 10.1378/chest.118.6.1680. PMID 11115458
- [Background] Kahn SR, Lim W, Dunn AS, Cushman M, Dentali F, Akl EA, Cook DJ, Balekian AA, Klein RC, Le H, Schulman S, Murad MH. Prevention of VTE in nonsurgical patients: Antithrombotic Therapy and Prevention of Thrombosis, 9th ed: American College of Chest Physicians Evidence-Based Clinical Practice Guidelines. Chest. 2012 Feb;141(2 Suppl):e195S-e226S. doi: 10.1378/chest.11-2296. PMID 22315261
- [Background] Office of the Surgeon General (US); National Heart, Lung, and Blood Institute (US). The Surgeon General's Call to Action to Prevent Deep Vein Thrombosis and Pulmonary Embolism. Rockville (MD): Office of the Surgeon General (US); 2008. Available from http://www.ncbi.nlm.nih.gov/books/NBK44178/ PMID 20669525
- [Background] Parikh AM, Spencer FA, Lessard D, Emery C, Baylin A, Linkletter C, Goldberg RJ. Venous thromboembolism in patients with reduced estimated GFR: a population-based perspective. Am J Kidney Dis. 2011 Nov;58(5):746-55. doi: 10.1053/j.ajkd.2011.06.021. Epub 2011 Aug 27. PMID 21872977
- [Background] Pavord S, Myers B. Bleeding and thrombotic complications of kidney disease. Blood Rev. 2011 Nov;25(6):271-8. doi: 10.1016/j.blre.2011.07.001. Epub 2011 Aug 26. PMID 21872374
- [Background] Bottger B, Wehling M, Bauersachs RM, Amann S, Schuchert A, Reinhold C, Kumpers P, Wilke T. Prevalence of renal insufficiency in hospitalised patients with venous thromboembolic events: a retrospective analysis based on 6,725 VTE patients. Thromb Res. 2014 Nov;134(5):1014-9. doi: 10.1016/j.thromres.2014.09.003. Epub 2014 Sep 9. PMID 25263017
- [Background] Cook D, Arabi Y, Ferguson N, Heels-Ansdell D, Freitag A, McDonald E, Clarke F, Keenan S, Pagliarello G, Plaxton W, Herridge M, Karachi T, Vallance S, Cade J, Crozier T, Alves da Silva S, Costa Filho R, Brandao N, Watpool I, McArdle T, Hollinger G, Mandourah Y, Al-Hazmi M, Zytaruk N, Adhikari NK; PROTECT Research Coordinators; PROTECT Investigators; Canadian Critical Care Trials Group; Australian and New Zealand Intensive Care Society Clinical Trials Group. Physicians declining patient enrollment in a critical care trial: a case study in thromboprophylaxis. Intensive Care Med. 2013 Dec;39(12):2115-25. doi: 10.1007/s00134-013-3074-x. PMID 24022796
- [Background] PROTECT Investigators for the Canadian Critical Care Trials Group and the Australian and New Zealand Intensive Care Society Clinical Trials Group; Cook D, Meade M, Guyatt G, Walter S, Heels-Ansdell D, Warkentin TE, Zytaruk N, Crowther M, Geerts W, Cooper DJ, Vallance S, Qushmaq I, Rocha M, Berwanger O, Vlahakis NE. Dalteparin versus unfractionated heparin in critically ill patients. N Engl J Med. 2011 Apr 7;364(14):1305-14. doi: 10.1056/NEJMoa1014475. Epub 2011 Mar 22. PMID 21417952
- [Background] Folsom AR, Lutsey PL, Astor BC, Wattanakit K, Heckbert SR, Cushman M; Atherosclerosis Risk in Communities Study. Chronic kidney disease and venous thromboembolism: a prospective study. Nephrol Dial Transplant. 2010 Oct;25(10):3296-301. doi: 10.1093/ndt/gfq179. Epub 2010 Mar 29. PMID 20353958
- [Background] Wattanakit K, Cushman M. Chronic kidney disease and venous thromboembolism: epidemiology and mechanisms. Curr Opin Pulm Med. 2009 Sep;15(5):408-12. doi: 10.1097/MCP.0b013e32832ee371. PMID 19561505
- [Background] Christiansen CF, Schmidt M, Lamberg AL, Horvath-Puho E, Baron JA, Jespersen B, Sorensen HT. Kidney disease and risk of venous thromboembolism: a nationwide population-based case-control study. J Thromb Haemost. 2014 Sep;12(9):1449-54. doi: 10.1111/jth.12652. Epub 2014 Jul 29. PMID 25040558
- [Background] Ocak G, Vossen CY, Verduijn M, Dekker FW, Rosendaal FR, Cannegieter SC, Lijfering WM. Risk of venous thrombosis in patients with major illnesses: results from the MEGA study. J Thromb Haemost. 2013 Jan;11(1):116-23. doi: 10.1111/jth.12043. PMID 23106832
- [Background] Kumar G, Sakhuja A, Taneja A, Majumdar T, Patel J, Whittle J, Nanchal R; Milwaukee Initiative in Critical Care Outcomes Research (MICCOR) Group of Investigators. Pulmonary embolism in patients with CKD and ESRD. Clin J Am Soc Nephrol. 2012 Oct;7(10):1584-90. doi: 10.2215/CJN.00250112. Epub 2012 Jul 26. PMID 22837271
- [Background] Fanikos J, Stevens LA, Labreche M, Piazza G, Catapane E, Novack L, Goldhaber SZ. Adherence to pharmacological thromboprophylaxis orders in hospitalized patients. Am J Med. 2010 Jun;123(6):536-41. doi: 10.1016/j.amjmed.2009.11.017. PMID 20569760
- [Background] Garcia DA, Baglin TP, Weitz JI, Samama MM. Parenteral anticoagulants: Antithrombotic Therapy and Prevention of Thrombosis, 9th ed: American College of Chest Physicians Evidence-Based Clinical Practice Guidelines. Chest. 2012 Feb;141(2 Suppl):e24S-e43S. doi: 10.1378/chest.11-2291. PMID 22315264
- [Background] Alikhan R, Bedenis R, Cohen AT. Heparin for the prevention of venous thromboembolism in acutely ill medical patients (excluding stroke and myocardial infarction). Cochrane Database Syst Rev. 2014 May 7;2014(5):CD003747. doi: 10.1002/14651858.CD003747.pub4. PMID 24804622
- [Background] Wilbur K, Lynd LD, Sadatsafavi M. Low-molecular-weight heparin versus unfractionated heparin for prophylaxis of venous thromboembolism in medicine patients--a pharmacoeconomic analysis. Clin Appl Thromb Hemost. 2011 Oct;17(5):454-65. doi: 10.1177/1076029610376935. Epub 2010 Aug 10. PMID 20699258
- [Background] Shorr AF, Jackson WL, Weiss BM, Moores LK. Low-molecular weight heparin for deep vein thrombosis prophylaxis in hospitalized medical patients: results from a cost-effectiveness analysis. Blood Coagul Fibrinolysis. 2007 Jun;18(4):309-16. doi: 10.1097/MBC.0b013e328099af58. PMID 17473570
- [Background] Lim W, Dentali F, Eikelboom JW, Crowther MA. Meta-analysis: low-molecular-weight heparin and bleeding in patients with severe renal insufficiency. Ann Intern Med. 2006 May 2;144(9):673-84. doi: 10.7326/0003-4819-144-9-200605020-00011. PMID 16670137
- [Background] Atiq F, van den Bemt PM, Leebeek FW, van Gelder T, Versmissen J. A systematic review on the accumulation of prophylactic dosages of low-molecular-weight heparins (LMWHs) in patients with renal insufficiency. Eur J Clin Pharmacol. 2015 Aug;71(8):921-9. doi: 10.1007/s00228-015-1880-5. Epub 2015 Jun 14. PMID 26071276
- [Background] Johansen KB, Balchen T. Tinzaparin and other low-molecular-weight heparins: what is the evidence for differential dependence on renal clearance? Exp Hematol Oncol. 2013 Aug 8;2:21. doi: 10.1186/2162-3619-2-21. eCollection 2013. PMID 23927414
- [Background] Mahe I, Aghassarian M, Drouet L, Bal Dit-Sollier C, Lacut K, Heilmann JJ, Mottier D, Bergmann JF. Tinzaparin and enoxaparin given at prophylactic dose for eight days in medical elderly patients with impaired renal function: a comparative pharmacokinetic study. Thromb Haemost. 2007 Apr;97(4):581-6. PMID 17393021
- [Background] Siguret V, Gouin-Thibault I, Pautas E, Leizorovicz A. No accumulation of the peak anti-factor Xa activity of tinzaparin in elderly patients with moderate-to-severe renal impairment: the IRIS substudy. J Thromb Haemost. 2011 Oct;9(10):1966-72. doi: 10.1111/j.1538-7836.2011.04458.x. PMID 21819539
- [Background] Douketis J, Cook D, Meade M, Guyatt G, Geerts W, Skrobik Y, Albert M, Granton J, Hebert P, Pagliarello G, Marshall J, Fowler R, Freitag A, Rabbat C, Anderson D, Zytaruk N, Heels-Ansdell D, Crowther M; Canadian Critical Care Trials Group. Prophylaxis against deep vein thrombosis in critically ill patients with severe renal insufficiency with the low-molecular-weight heparin dalteparin: an assessment of safety and pharmacodynamics: the DIRECT study. Arch Intern Med. 2008 Sep 8;168(16):1805-12. doi: 10.1001/archinte.168.16.1805. PMID 18779469
- [Background] Cook DJ, Rocker G, Meade M, Guyatt G, Geerts W, Anderson D, Skrobik Y, Hebert P, Albert M, Cooper J, Bates S, Caco C, Finfer S, Fowler R, Freitag A, Granton J, Jones G, Langevin S, Mehta S, Pagliarello G, Poirier G, Rabbat C, Schiff D, Griffith L, Crowther M; PROTECT Investigators; Canadian Critical Care Trials Group. Prophylaxis of Thromboembolism in Critical Care (PROTECT) Trial: a pilot study. J Crit Care. 2005 Dec;20(4):364-72. doi: 10.1016/j.jcrc.2005.09.010. PMID 16310609
- [Background] Mariani AW, Pego-Fernandes PM. Observational studies: why are they so important? Sao Paulo Med J. 2014;132(1):1-2. doi: 10.1590/1516-3180.2014.1321784. No abstract available. PMID 24474072
- [Background] Hainer JW, Sherrard DJ, Swan SK, Barrett JS, Assaid CA, Fossler MJ, Cox DS, Williams RM, Pittenger AL, Stephenson CA, Hua TA. Intravenous and subcutaneous weight-based dosing of the low molecular weight heparin tinzaparin (Innohep) in end-stage renal disease patients undergoing chronic hemodialysis. Am J Kidney Dis. 2002 Sep;40(3):531-8. doi: 10.1053/ajkd.2002.34911. PMID 12200805
- [Background] Sanderink GJ, Guimart CG, Ozoux ML, Jariwala NU, Shukla UA, Boutouyrie BX. Pharmacokinetics and pharmacodynamics of the prophylactic dose of enoxaparin once daily over 4 days in patients with renal impairment. Thromb Res. 2002 Feb 1;105(3):225-31. doi: 10.1016/s0049-3848(02)00031-2. PMID 11927128
- [Background] Schmid P, Brodmann D, Odermatt Y, Fischer AG, Wuillemin WA. Study of bioaccumulation of dalteparin at a therapeutic dose in patients with renal insufficiency. J Thromb Haemost. 2009 Oct;7(10):1629-32. doi: 10.1111/j.1538-7836.2009.03556.x. Epub 2009 Jul 17. PMID 19624460
- [Background] Li L, Li X, Xu L, Sheng Y, Huang J, Zheng Q. Systematic evaluation of dose accumulation studies in clinical pharmacokinetics. Curr Drug Metab. 2013 Jun;14(5):605-15. doi: 10.2174/13892002113149990002. PMID 23701162
- [Background] Michels WM, Grootendorst DC, Verduijn M, Elliott EG, Dekker FW, Krediet RT. Performance of the Cockcroft-Gault, MDRD, and new CKD-EPI formulas in relation to GFR, age, and body size. Clin J Am Soc Nephrol. 2010 Jun;5(6):1003-9. doi: 10.2215/CJN.06870909. Epub 2010 Mar 18. PMID 20299365
- [Background] van Veen JJ, Gatt A, Makris M. Thrombin generation testing in routine clinical practice: are we there yet? Br J Haematol. 2008 Sep;142(6):889-903. doi: 10.1111/j.1365-2141.2008.07267.x. Epub 2008 Jun 28. PMID 18564356
- [Background] Leizorovicz A, Bara L, Samama MM, Haugh MC. Factor Xa inhibition: correlation between the plasma levels of anti-Xa activity and occurrence of thrombosis and haemorrhage. Haemostasis. 1993 Mar;23 Suppl 1:89-98. doi: 10.1159/000216915. PMID 8388357
- [Background] Ignjatovic V, Summerhayes R, Gan A, Than J, Chan A, Cochrane A, Bennett M, Horton S, Shann F, Lane G, Ross-Smith M, Monagle P. Monitoring Unfractionated Heparin (UFH) therapy: which Anti-Factor Xa assay is appropriate? Thromb Res. 2007;120(3):347-51. doi: 10.1016/j.thromres.2006.10.006. Epub 2006 Nov 21. PMID 17118432
- [Background] Crowther M, Lim W. Low molecular weight heparin and bleeding in patients with chronic renal failure. Curr Opin Pulm Med. 2007 Sep;13(5):409-13. doi: 10.1097/MCP.0b013e328216430d. PMID 17940486
- [Background] Bara L, Leizorovicz A, Picolet H, Samama M. Correlation between anti-Xa and occurrence of thrombosis and haemorrhage in post-surgical patients treated with either Logiparin (LMWH) or unfractionated heparin. Post-surgery Logiparin Study Group. Thromb Res. 1992 Mar 1;65(4-5):641-50. doi: 10.1016/0049-3848(92)90213-t. PMID 1319619
- [Background] Atiq F, van den Bemt PM, Leebeek FW, van Gelder T, Versmissen J. No accumulation of a prophylactic dose of nadroparin in moderate renal insufficiency. Neth J Med. 2015 Oct;73(8):373-8. PMID 26478547
- [Background] Dobromirski M, Cohen AT. How I manage venous thromboembolism risk in hospitalized medical patients. Blood. 2012 Aug 23;120(8):1562-9. doi: 10.1182/blood-2012-03-378901. Epub 2012 Jun 15. PMID 22705598